CLINICAL TRIAL: NCT06241456
Title: A Phase 1 Study of FT825/ONO-8250, an Off-the-Shelf CAR T-Cell Therapy, With or Without Monoclonal Antibodies, in HER2-Positive or Other Advanced Solid Tumors
Brief Title: FT825/ONO-8250, an Off-the-Shelf, HER2 CAR-T, With or Without Monoclonal Antibodies in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT825-101
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Bendamustine Hydrochloride; Docetaxel; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A: FT825 (Experimental): Participants with advanced HER2-expressing solid tumors receive FT825 following chemotherapy in Cycle 1 (each cycle is approximately 61 days). Based on the safety, tolerability, and radiographically confirmed clinical benefit to treatment in Cycle 1, participants may be considered for an additional treatment cycle (Cycle 2 retreatment).
  Interventions: Drug: FT825; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Bendamustine; Drug: Docetaxel; Drug: Cisplatin
- Regimen B: FT825 + Cetuximab (Experimental): Participants with advanced epidermal growth factor receptor (EGFR)-expressing solid tumors receive FT825 in combination with cetuximab following chemotherapy in Cycle 1 (each cycle is approximately 61 days). Based on the safety, tolerability, and radiographically confirmed clinical benefit to treatment in Cycle 1, participants may be considered for an additional treatment cycle (Cycle 2 retreatment).
  Interventions: Drug: FT825; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Bendamustine; Drug: Docetaxel; Drug: Cisplatin; Drug: Cetuximab

INTERVENTIONS:
Drug: FT825 — FT825 will be administered as an intravenous (IV) infusion at planned dose levels.
  Other Names: ONO-8250
Drug: Fludarabine — Fludarabine will be administered as an IV infusion at planned dose levels.
  Other Names: FLUDARA
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an IV infusion at planned dose levels.
Drug: Bendamustine — Bendamustine will be administered as an IV infusion at planned dose levels.
Drug: Docetaxel — Docetaxel will be administered as an IV infusion at planned dose levels.
Drug: Cisplatin — Cisplatin will be administered as an IV infusion at planned dose levels.
Drug: Cetuximab — Cetuximab will be administered as an IV infusion at planned dose levels.
  Arms: Regimen B: FT825 + Cetuximab

SUMMARY:
This is a phase 1 study designed to evaluate the safety, tolerability, and antitumor activity of FT825 (also known as ONO-8250) with or without monoclonal antibody therapy following chemotherapy in participants with advanced human epidermal growth factor receptor 2 (HER2)-positive or other advanced solid tumors. The study will consist of a dose-escalation stage, followed by an expansion stage to further evaluate the safety and activity of FT825 in indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological or cytologically confirmed locally advanced or metastatic cancer that meets protocol-defined criteria
* Disease that is not amenable to curative therapy, with prior therapies defined by specific tumor types
* Contraceptive use by women and men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Presence of measurable disease by RECIST, v1.1 assessed within 28 days prior to start of first study intervention
* Anticipated life expectancy of at least 3 months

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Evidence of inadequate organ function
* Clinically significant cardiovascular disease
* Known active central nervous system (CNS) involvement by malignancy
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions within 2 years prior to study enrollment
* Active bacterial, fungal, or viral infections
* Prior receipt of chimeric antigen receptor (CAR) T-cell therapy, other cellular therapy, or a FATE investigational human induced pluripotent stem cell (iPSC) product
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out based on imaging at screening
* Any history of Grade ≥3 immune-related AE or Grade ≥2 eye toxicity attributed to prior cancer immunotherapy, other than endocrinopathy managed with replacement therapy or asymptomatic elevation of serum amylase or lipase
* Active or history of autoimmune disease or immune deficiency
* Receipt of an allograft organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2044-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | Up to approximately 29 days
  The number of participants with DLTs will be reported.
Number of participants with treatment-emergent adverse events (TEAEs) | Up to approximately 2 years
  The number of participants with TEAEs will be reported.
Severity of AEs | Up to approximately 2 years
  Severity of AEs will be determined according to appropriate rating scales for the type of event reported.

SECONDARY OUTCOMES:
Investigator-Assessed Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is the proportion of participants who achieve partial response (PR) or complete response (CR) per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST, v.1.1).
Investigator-Assessed Duration of Response (DOR) | Up to approximately 2 years
  DOR is the duration from the first occurrence of a documented objective response of either PR or CR until the time of disease progression, or death from any cause, whichever occurs first, per RECIST, v.1.1.
Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is the time from first dose of study intervention to disease progression, or to the day of death for any reason, whichever occurs first, per RECIST, v.1.1.
Overall Survival (OS) | Up to approximately 2 years
  OS defined as the time from first dose of study intervention to death from any cause.
Plasma Concentration of FT825 | At designated time points up to approximately 56 days
  The plasma concentration of FT825 will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Fate Therapeutics
Locations (14):
- United States (14):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Yale New Haven Hospital - Yale Cancer Center, New Haven, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oncology Hematology Care Clinial Trials, Cincinnati, Ohio
  - Ohio State University - Comprehensive Cancer Center, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute (SCRI) - Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas